CLINICAL TRIAL: NCT03193580
Title: Accelerating Motor Learning in Pediatrics
Acronym: AMPED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Adam Kirton, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: REB16-2474
Record Dates: First submitted 2017-05-05; First posted 2017-06-21 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Healthy; Pediatrics
Keywords: Anodal Stimulation Transcranial Direct Current Stimulation; High-Definition Transcranial Direct Current Stimulation; tDCS; Non-invasive brain stimulation; Pediatrics

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of three groups (sham, tDCS, HD-tDCS) throughout the duration of the study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anodal Conventional tDCS (Experimental): The intervention will be anodal conventional tDCS. Anodal tDCS: 30 second ramp up to 1milliamp, 20 minute current hold at 1milliamp, 30 second ramp down to 0 milliamp. Anode positioned over the right primary motor cortex, and the cathode over the contralateral supraorbital area.
  Interventions: Device: Anodal Conventional tDCS
- Anodal High Definition tDCS (Experimental): The intervention will be anodal high definition-tDCS. Anodal HD-tDCS: 30 second ramp up to 1milliamp, 20 minute current hold at 1milliamp, 30 second ramp down to 0milliamp. Anode entered over the right primary motor cortex, and four cathodes placed in a ring formation surrounding the anode.
  Interventions: Device: Anodal High Definition tDCS
- Sham tDCS (Sham Comparator): Sham subjects will undergo exactly the same anodal conventional tDCS protocol as outlined above. This includes the initial stimulation sequence of ramp up of 30 seconds, generating the initial transient scalp sensations identical to the treatment group. The stimulator will be programmed by the technologist after 120 seconds of stimulation to automatically ramp down to 0milliamp over 30 seconds.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Anodal Conventional tDCS — tDCS will be applied for 20 minutes at 1milliamp while participants are performing a fine motor task. The current will be set at 1milliamp, stimulation will be ramped up over 30 seconds and ramped down over 30 seconds.
  Other Names: Direct-current stimulator (Soterix)
  Arms: Anodal Conventional tDCS
Device: Anodal High Definition tDCS — HD-tDCS will be applied for 20 minutes at 1milliamp while participants are performing a fine motor task. The current will be set at 1milliamp, stimulation will be ramped up over 30 seconds and ramped down over 30 seconds.
  Other Names: Direct-current stimulator (Soterix)
  Arms: Anodal High Definition tDCS
Device: Sham tDCS — tDCS will be applied for 1 minutes at 1milliamp while participants are performing a fine motor task. The current will be set at 1milliamp, stimulation will be ramped up over 30 seconds and ramped down over 30 seconds.
  Other Names: Direct-current stimulator (Soterix)
  Arms: Sham tDCS

SUMMARY:
Non-invasive brain stimulation can both study and potentially treat neurological disorders. Transcranial direct-current stimulation (tDCS) is an emerging safe and tolerability form of stimulation and has been used increasingly over the last decade.

The purpose of this research is to see if two different types of tDCS can improve motor function in healthy children. tDCS has been shown to safely enhance hand motor function in healthy adults, and those that have suffered stroke and other conditions. Recently the investigators demonstrated that tDCS may enhance hand motor function in healthy children, however, how it does so is unknown. In addition to assessing changes in motor function when tDCS is given during motor skill training, the investigators will perform various tests before and after stimulation to understand the changes that happen in the brain accompanying motor skill learning and brain stimulation.

The investigators hypothesize that there will be an accelerated acquisition of motor skill, when training is paired with conventional anodal tDCS, HD-tDCS, or sham tDCS.

DETAILED DESCRIPTION:
Background & rationale: Plasticity may be enhanced in the developing brain but mechanisms are poorly understood. Brain stimulation technologies such as transcranial direct-current stimulation (tDCS) modulate motor cortex excitability and plasticity. Studies by our group and others suggest that neuromodulation trials with tDCS are both safe and feasible in children. Recently the investigators demonstrated that conventional tDCS can enhance motor learning in healthy children. Additionally, recent advances in high-definition tDCS (HD-tDCS) have presented an opportunity to focally stimulate regions of the brain. HD-tDCS has not been investigated to date in children.

Establishing an ability of tDCS to enhance motor learning has therapeutic implications for children with motor disabilities. Perinatal stroke is the leading cause of hemiparetic cerebral palsy and most survivors suffer lifelong physical disability. Emerging models from our lab and others have defined central therapeutic targets whereby brain stimulation may enhance motor learning and function. Understand the effects of tDCS on motor learning, and it's underlying changes within the brain, is essential to advancing such interventions.

Research question & objectives: Here the investigators propose to characterize the effects of tDCS on motor learning in healthy children. The primary objective of this study is to determine changes in acquisition of motor skill, when training is paired with conventional anodal tDCS, HD-tDCS, or sham tDCS. Multiple secondary objectives will describe biochemical and sensorimotor changes in the brain that take place during motor learning paired with tDCS. Secondary objectives will also assess the safety of HD- tDCS in healthy children.

Ethics: This study has been approved by the University of Calgary Research Ethics Board.

Design: Randomized, double blind, sham-controlled trial to evaluate the ability of tDCS and HD-tDCS to enhance motor learning.

Methods: Children will be recruited through the Healthy Infants and Children Clinical Research Program.

The training task will consists of performing the Purdue Pegboard Test (PPTL) with their left hand. This simple motor learning task is a well-validated task for complex, functionally relevant motor learning. The PPTL has demonstrated good sensitivity to change in both healthy and disease motor learning studies in adults and school-aged children. The PPTL will be performed over five consecutive days to monitor motor learning.

Children will attend the Alberta Children's Hospital Non-Invasive Brain Stimulation Laboratory. Subjects will be randomized to one of three stimulation groups (sham tDCS, conventional anodal tDCS, HD-tDCS). Baseline measures will be performed, including: magnetic resonance neuroimaging (anatomical imaging, functional neuroimaging and magnetic resonance spectroscopy), transcranial magnetic stimulation neurophysiology (motor mapping of the left and right motor cortex), sensorimotor functional changes assessed using the Kinesiological Instrument for Normal and Altered Reaching Movements (KINARM; arm positioning matching, kinesthesia, visually guided reaching, and object hit task), motor function changes (PPT, Jebsen-Taylor Test, Serial Reaction Time Task), and sensory discrimination measures (amplitude discrimination, temporal order judgment, temporal order judgment task, duration discrimination task, duration discrimination with confound, and single site adaptation task.

Following baseline measures, subjects will be seating in a comfortable chair with the PPTL test in front of them on a table. Participant randomized to sham or conventional anodal tDCS will be fitted with two 25cm2 electrodes (anode over the right primary motor cortex, cathode over the contralateral supraorbital area) or an EEG cap containing four small circular electrode (HD-tDCS, 1 anode centered over the right primary motor cortex, 4 cathodes surround the anode in a ring-like fashion). Three pre-intervention trials of the PPTL will be performed. All subjects will then have the tDCS ramped up to 1milliamp over 45 seconds. After 120 seconds the current will either be ramped down to 0milliamp (sham tDCS) or continue for a total of 20 minutes. The PPTL will be performed 5, 10, and 15 minutes following stimulation commencement, and after stimulation has ended (3 repetitions per time point). A tDCS safety and tolerability questionnaire will then be completed.

The same tDCS-treatment, PPTL training and safety and tolerability questionnaires will be performed over the next three consecutive days. On study day 5 participants will again repeat PPTL training paired with tDCS-treatment. Following tDCS and PPTL training, magnetic resonance neuroimaging, transcranial magnetic stimulation neurophysiology, sensorimotor functional changes, motor function changes, and sensory discrimination measures will be repeated to assess changes induced by motor learning and tDCS.

Participants will return six weeks following training, where magnetic resonance neuroimaging, transcranial magnetic stimulation neurophysiology, sensorimotor functional changes, motor function changes, and sensory discrimination measures will be repeated to assess long-term changes.

Data analysis: All outcome variables will be compared across the three intervention groups (sham tDCS, conventional tDCS, HD- tDCS) using a two-way repeated measures ANOVA with appropriate post-hoc analysis. The repeated measures ANOVA will distinguish the influence of intervention (stimulation type) and time (baseline, post-training, 1 month post- training). Pearson's correlations will be performed between the primary outcome measure and secondary outcome measures. Secondary statistical analysis will be performed as warranted.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-18 years
* Right-handed
* Normal development
* No neuropsychiatric disorders, neuropsychotropic medications, or chronic medical conditions
* Informed consent/assent

Exclusion Criteria:

* Implanted electrical devices, including (but not limited to) cardiac pacemakers.
* Metallic implants or irremovable metal objects
* Pregnant females or females who may be pregnant.
* Braces or upper teeth wires.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Left Hand Purdue Pegboard Test Score | Baseline and immediately post-training on day 5
  A "baseline" trial will be performed. Each day they will do 15 repetitions for 5 consecutive days. On the fifth day, they will do a post training trial consisting of 3 repetitions.

SECONDARY OUTCOMES:
Percent change in metabolic markers | Baseline, post-training on day 5, and 6 weeks following training
  Metabolic markers including GABA and glutamate will be assessed using Magnetic Resonance Spectroscopy (MRS). An MRS will be performed at baseline, on day 5 post-training, and at the 6 week follow-up.
Raw change in functional motor activations | Baseline, post-training on day 5, and 6 weeks following training
  Measures of functional motor activity will be assessed using Functional Magnetic Resonance Imaging (MRI). Finger-tapping task will be performed in the MRI scanner. An MRI will be performed at baseline, on day 5 post-training, and at the 6 week follow-up.
Raw change in robotic sensorimotor measures | Baseline, post-training on day 5, and 6 weeks following training
  The Kinesiological Instrument for Normal and Altered Reaching Movements (KINARM). The raw change in measures of proprioception, kinesthesia, visually-guided reaching, and object hit tasks will be measured. On the fifth day, the participants will do a post-training trial.
Raw change in vibro-tactile sensory measures | Baseline, post-training on day 5, and 6 weeks following training
  The raw change of the Brain Gauge vibro-tactile sensory assessment score will be measured. On the fifth day, the participants will do a post-training trial.
Raw change in size of transcranial magnetic stimulation (TMS) motor maps | Baseline, post-training on day 5, and 6 weeks following training
  The raw change in TMS-measured motor evoked potential amplitude (Microvolts,uV) and neurophysiological changes in motor evoked potential size (Microvolts,uV). On the fifth day, the participants will do a post-training trial. Six weeks following the end of training, the participants will perform the task.
Raw change in motor function tasks - Serial Reaction Time test | Baseline, post-training on day 5, and 6 weeks following training
  Raw change in score on the Serial Reaction Time test. A "baseline" trial will be performed. On the fifth day, the participants will do a post-training trial. All tasks are measured in milliseconds. Six weeks following the end of training, the participants will perform the task.
Raw change in motor function tasks - Jebsen-Taylor test | Baseline, post-training on day 5, and 6 weeks following training
  Raw change in score on the Jebsen-Taylor test. A "baseline" trial will be performed. All measures are measured in seconds. On the fifth day, the participants will do a post-training trial. Six weeks following the end of training, the participants will perform the task.
Raw change in motor function tasks - Purdue Pegboard test | Baseline, post-training on day 5, and 6 weeks following training
  Raw change in score on the Purdue Pegboard Test for the left, right, and both hands. A "baseline" trial will be performed. The average number of pegs places will be measured. On the fifth day, they will do a post training trial consisting of 3 repetitions for the left, right, and both hands trials. Six weeks following the end of training, the participants will perform 3 repetitions for the left, right and both hands trials.

OTHER OUTCOMES:
Tolerability questionnaire | Baseline, following stimulation daily, and 6 weeks following training
  TMS and tDCS safety and tolerability. The questionnaire will be filled out after daily stimulation and at follow-up at 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Kirton, MD, MSc, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - Alberta Childrens Hospital, Calgary, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirton A, Ciechanski P, Zewdie E, Andersen J, Nettel-Aguirre A, Carlson H, Carsolio L, Herrero M, Quigley J, Mineyko A, Hodge J, Hill M. Transcranial direct current stimulation for children with perinatal stroke and hemiparesis. Neurology. 2017 Jan 17;88(3):259-267. doi: 10.1212/WNL.0000000000003518. Epub 2016 Dec 7. PMID 27927938
- [Background] Ciechanski P, Kirton A. Transcranial Direct-Current Stimulation Can Enhance Motor Learning in Children. Cereb Cortex. 2017 May 1;27(5):2758-2767. doi: 10.1093/cercor/bhw114. PMID 27166171
- [Background] Kuczynski AM, Semrau JA, Kirton A, Dukelow SP. Kinesthetic deficits after perinatal stroke: robotic measurement in hemiparetic children. J Neuroeng Rehabil. 2017 Feb 15;14(1):13. doi: 10.1186/s12984-017-0221-6. PMID 28202036
- [Background] Kuczynski AM, Dukelow SP, Semrau JA, Kirton A. Robotic Quantification of Position Sense in Children With Perinatal Stroke. Neurorehabil Neural Repair. 2016 Sep;30(8):762-72. doi: 10.1177/1545968315624781. Epub 2016 Jan 7. PMID 26747126
- [Derived] Cole L, Giuffre A, Ciechanski P, Carlson HL, Zewdie E, Kuo HC, Kirton A. Effects of High-Definition and Conventional Transcranial Direct-Current Stimulation on Motor Learning in Children. Front Neurosci. 2018 Oct 31;12:787. doi: 10.3389/fnins.2018.00787. eCollection 2018. PMID 30429768
- See also: Program website — http://www.perinatalstroke.ca